CLINICAL TRIAL: NCT03633422
Title: Evaluation of Stroke Patient Screening in an Acute Stroke Setting
Brief Title: Evaluation of Stroke Patient Screening
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2017-00844
Record Dates: First submitted 2018-07-24; First posted 2018-08-16 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Stroke, Acute
Keywords: Rehabilitation; Screening; Enrollment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and Rationale:

Traditionally, stroke rehabilitation studies have been performed in stroke patients beyond the first one to three months poststroke [Stinear et al. 2013; Veerbeek et al. 2014]. Acknowledging that early stroke rehabilitation should be initiated soon after stroke onset to optimize stroke outcomes, it is has been stressed that stroke rehabilitation trials should be initiated within the first month [Stinear 2013].

Early stroke rehabilitation trials face difficulties regarding patient recruitment with corresponding low enrollment rates [AVERT 2015; Winters 2015]. Explanations are for example priority given to (sub)acute medical interventions, highly dynamic situation at a stroke unit, and a more rapid change in patients' abilities when compared to patients in later stages poststroke. With the low enrollment rates (~7%), the generalizability of study results is questionable.

Participant screening methods and procedures for research eligibility are part of the patient selection and recruitment process in clinical trials. However, no information is available regarding screening procedures and methods for these early initiated stroke rehabilitation trials, including reasons for not enrolling patients. This knowledge is essential to improve screening procedures and methods, in order to optimize patient enrollment and with that, increase the generalizability of study results.

Objective:

The objective of this project is to evaluate screening methods and procedures for stroke rehabilitation research.

Study Design:

Observational study

DETAILED DESCRIPTION:
Objective:

The objective of this project is to evaluate screening methods and procedures for stroke rehabilitation research in the Department of Neurology, University Hospital Zurich.

Outcome:

Enrollment rates (defined as the number of patients enrolled per month of recruitment), reasons for non-enrollment, and estimated costs for screening for early stroke rehabilitation studies.

Study Design:

Observational study

ELIGIBILITY:
Inclusion Criteria:

* First-ever unilateral ischemic stroke <48 hours, confirmed by MRI-DWI and/or CT
* Age 18 years or older
* Able to follow one-staged commands
* NIHSS arm score ≥1
* Informed consent after participants' information

Exclusion Criteria:

* Modified Rankin Scale score >2 before stroke
* Neurological or other diseases affecting the upper limb(s) before stroke
* Intravenous line in the upper limb(s) which limits assessment
* Contra-indications on ethical grounds
* Expected or known non-compliance to participate in the observational study, severe drug or/and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stroke patients admitted to the University Hospital Zurich, Department of Neurology, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 845 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Reasons why participants are not eligible for an early rehabilitation trial | 1 Day
  The reasons for non-enrollment will be measured by counting, based on the inclusion and exclusion criteria of the aRISE study

SECONDARY OUTCOMES:
Enrolment rate | 1 Month
  Defined as the number of patients enrolled per month of screening
Estimated personnel expenses in Swiss Francs for screening | 1 Month
  Swiss Francs associated with screening in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Zürcher RehaZentrum Wald, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AVERT Trial Collaboration group. Efficacy and safety of very early mobilisation within 24 h of stroke onset (AVERT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):46-55. doi: 10.1016/S0140-6736(15)60690-0. Epub 2015 Apr 16. PMID 25892679
- [Background] Stinear C, Ackerley S, Byblow W. Rehabilitation is initiated early after stroke, but most motor rehabilitation trials are not: a systematic review. Stroke. 2013 Jul;44(7):2039-45. doi: 10.1161/STROKEAHA.113.000968. Epub 2013 May 28. No abstract available. PMID 23715959
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Winters C, van Wegen EE, Daffertshofer A, Kwakkel G. Generalizability of the Proportional Recovery Model for the Upper Extremity After an Ischemic Stroke. Neurorehabil Neural Repair. 2015 Aug;29(7):614-22. doi: 10.1177/1545968314562115. Epub 2014 Dec 11. PMID 25505223
- [Result] Held JPO, van Duinen J, Luft AR, Veerbeek JM. Eligibility Screening for an Early Upper Limb Stroke Rehabilitation Study. Front Neurol. 2019 Jul 2;10:683. doi: 10.3389/fneur.2019.00683. eCollection 2019. PMID 31312170